CLINICAL TRIAL: NCT06187064
Title: Combination Primary Care and Prevention Services for Women Who Inject Drugs and Exchange Sex in Seattle, Washington
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Maria Corcorran, Assistant Professor, School of Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00015337; R34DA054588-01A1 (NIH)
Record Dates: First submitted 2023-12-05; First posted 2024-01-02 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Opioid Use Disorder; HIV Infections; Chlamydia; Gonorrhea; Syphilis; Trichomonas
Keywords: Women who inject drugs; Medications for opioid use disorder; HIV pre-exposure prophylaxis; Venue-based healthcare
MeSH Terms: conditions — Opioid-Related Disorders; HIV Infections; Chlamydia Infections; Gonorrhea; Syphilis; Trichomonas Infections

STUDY DESIGN:
Intervention Model Description: Pilot of novel care model for low-barrier care and adherence support for uptake and sustained use of biomedical HIV prevention and medications for opioid use disorder for women who inject drugs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study cohort (Other): The investigators will enroll 50 female-identifying people who present to the clinical van for care and follow them for 6 months. The investigators will assess uptake of PrEP and buprenorphine; POC STI testing and treatment completion rates; sustained use of PrEP and buprenorphine at months 3 and 6 (n=50). The investigators will conduct surveys to assess and characterize the acceptability and feasibility of venue-based primary and HIV prevention care among women who inject drugs (WWID).
  Interventions: Other: Mobile Van Clinic

INTERVENTIONS:
Other: Mobile Van Clinic — The investigators will implement a pilot clinic one evening per week, with the primary goal of measuring a community-based extension of SHE Clinic's impact on uptake and sustained use of HIV pre-exposure prophylaxis (PrEP) and medications for opioid use disorder (MOUD). The clinic will be dispatched with a driver, nurse, physician, and research assistant. The van clinic will be outfitted with space to obtain a confidential history and physical exam and include a space for sample collection. In addition to standard of care, the investigators will provide participants with rapid point-of-care HIV and STI testing, and HIV PrEP and MOUD counseling and prescriptions.

SUMMARY:
The investigators will implement a non-randomized observational clinical trial that will include a pop-up clinic for women who inject drugs (WWID) near venues for exchange sex and drug use in north Seattle. The pop-up clinic will be housed within a van and serve as a research extension of the SHE Clinic, a Harborview Medical Center run clinic for women who exchange sex and use drugs in north Seattle. Through the implementation of the pop-up clinic, the investigators will aim to assess:

1. The impact of the pop-up clinic on uptake and sustained use of HIV pre-exposure prophylaxis (PrEP) and medications for opioid use disorder (MOUD) among WWID.
2. The impact of point of care (POC) sexually transmitted infection (STI) testing on STI treatment completion rates.
3. The acceptability and feasibility of providing HIV prevention care for WWID and exchange sex in a pop-up van clinic.

DETAILED DESCRIPTION:
The investigators will implement a pilot clinic one evening per week, with the primary goal of measuring a community-based extension of SHE Clinic's impact on uptake and sustained use of HIV pre-exposure prophylaxis (PrEP) and medications for opioid use disorder (MOUD). The clinic will be dispatched with a driver, nurse, physician, and research assistant. The van clinic will be outfitted with space to obtain a confidential history and physical exam and include a space for sample collection. Similarly, the van clinic will be equipped with a WiFi hotspot with a laptop linked to University of Washington's electronic medical record (EMR) system for clinical documentation, orders, and referrals. In addition to standard of care, the investigators will provide participants with rapid point-of-care HIV and STI testing. All people presenting for a walk-in clinic visit who do not enroll will be offered laboratory-based testing and prescription medications, which are subject to insurance/billing, per standard of care. Women enrolled in the research study will be instructed on self-collection of vaginal swab specimens, which will be tested for C. trachomatis and N. gonorrhoeae using the 30-minute Binx Health rapid PCR platform. OSOM swabs for trichomonas will be placed into a sterile tube and processed on site with rapid testing kits (Sekisui Diagnostics) along with POC HIV and syphilis testing via finger prick (Chembio Diagnostic Systems). Any samples that cannot be tested using point-of-care methods will be transported to Harborview Medical Center laboratory following clinic sessions. Results will be delivered to participants, either immediately, via cell phone for lab-based tests or when a participant follows up at the mobile clinic or at SHE Clinic. STI treatment will be given per clinical guidelines.

Results will be noted in participants' EMR for improved continuity of care across the healthcare system. Study participants who return for results (or receive them via phone) and undergo appropriate treatment, if necessary. This novel venue-based clinic will be integrated within the larger University of Washington (UW) healthcare system, and necessary referrals will be made to UW facilities, including a large UW medical campus located two miles north of Aurora Commons. Participants not already registered in the UW system will receive a medical record number and clinical portions of study visits will be documented in EMR to improve overall continuity of care. Referrals for syringe services will similarly be made to a local syringe service program. Additional dedicated research activities taking place in this care model will include surveys and adherence monitoring via dried blood spot (DBS), as detailed below. Adherence support will be incorporated into this model using established evidence-based approaches in response to the analysis of formative qualitative work and recommendations of the community advisory board.

Clinical study visits will occur at enrollment, a follow-up study visit at month-3, and an exit visit at 6-months post-enrollment. For participants who are prescribed buprenorphine, additional brief refill visits will occur at monthly intervals. All assessments will occur during in-person visits in the pilot clinic. Each study visit will consist of a short survey, an eligibility assessment for oral PrEP and MOUD, standard clinical care, and biological sample collections (i.e., DBS sample collection for research only, self-collected vaginal swabs for point-of-care STI testing, and blood samples for blood born infection testing). To test the impact of this pilot clinic model on improving uptake and sustained use of HIV prevention services, the investigators will utilize medical record data and hair drug (buprenorphine and tenofovir) levels. Dried blood spot samples will be collected as a backup method to evaluate adherence. Prior to enrollment, participants will be asked to provide consent for participation in the study, review of EMR data, and review of pharmacy records. Consent will be collected using electronic data capture (REDCap) and participant data will be collected by medical record number (MRN) utilizing an EMR querying technology (Leaf) generated by the University of Washington as well as manual chart review. Participants meeting CDC eligibility criteria for PrEP will be counseled on HIV risk, offered HIV testing, and if negative and interested, oral PrEP will be prescribed per clinical guidelines. Additionally, participants with active self-reported use of opioids will be counseled on options for opioid use disorder treatment, and those interested in MOUD, will be provided with a prescription for buprenorphine-naloxone or buprenorphine, per clinical guidelines. Uptake of PrEP and buprenorphine will be measured by review of pharmacy and EMR records and will be defined by filling a prescription for PrEP or buprenorphine. The investigators will measure sustained use of PrEP and buprenorphine via tenofovir disoproxil fumarate (TDF) and buprenorphine levels in samples of 150 hairs. The investigators can simultaneously test for buprenorphine, fentanyl and tenofovir from the same specimen, and will measure these drug levels at 3- and 6- months to evaluate adherence to PrEP and buprenorphine. Additionally, dried blood spots (DBS) will be collected and archived to ensure that drug levels are collected during this study in the event there are any complications with hair testing.

At each visit, brief demographic and behavioral surveys will be administered to women enrolled in the study via tablets, with responses recorded in REDCap. At the end of each visit an additional survey assessing acceptability of venue-based care will be administered to each participant. Questions will be informed by the CFIR and designed to assess the acceptability and relative priority of venue-based primary and HIV prevention care among women seeking services. As part of an assessment of acceptability, questions will also focus on the perceived stigma associated with receipt of care at the pop-up van clinic near a venue for drug use and exchange sex. Following completion of the intervention, information on feasibility, implementation barriers and facilitators will be collected using semi-structured interviews with clinical staff to contextualize logistical and structural barriers faced by venue-based service delivery.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Female identifying
* Ever injected drugs
* Not known to have HIV
* Willing and able to provide informed consent to participate in the study

Exclusion Criteria:

* <18 years of age
* Never injected drugs
* Living with HIV
* Medical or psychological co-morbidities that prevent participation per study team assessment.
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female identifying
Enrollment: 50 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Evaluate uptake of PrEP and MOUD | 6 months
  Proportion of participants who initiate PrEP and/or MOUD

OTHER OUTCOMES:
Evaluate sustained use of PrEP and MOUD | 6 months
  Proportion of participants who achieve continued use of PrEP and/or MOUD
Evaluate treatment completion rate after POC STI testing | 6 months
  Proportion of participants who complete STI treatment following a reactive/positive STI test
Evaluate testing time to completion after POC STI testing | 6 months
  Time from reactive/positive STI test to completion of STI treatment
Assess acceptability of pilot community-based care model | 6 months
  Proportion of participants who agree that care model is safe and that their health improved getting care from a mobile clinic
Assess acceptability of POC STI testing at community-based site | 6 months
  Proportion of participants who agree that they felt comfortable getting and/or prefer POC STI testing

CONTACTS AND LOCATIONS:
Overall Officials: Maria Corcorran, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT06187064/Prot_000.pdf